CLINICAL TRIAL: NCT03604770
Title: Caloric Intake and Ovarian Reserve
Status: Withdrawn | Type: Observational
Why Stopped: Due to lack of enrollment.
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 17028
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Infertility, Female
Keywords: Caloric Intake; Anti-mullerian hormone (AMH); Antral follicles (AFC); Infertility; Fertility; Diet; Ovarian Reserve; Obesity; Nutrition
MeSH Terms: conditions — Infertility, Female; Infertility; Obesity | interventions — Surveys and Questionnaires; Diet Records

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women seeking fertility treatment: Women aged 18-45 who are seeking fertility treatment at Bethesda Fertility Center will be provided a survey and food diary to complete.
  Interventions: Other: Survey & Food Diary

INTERVENTIONS:
Other: Survey & Food Diary — Patients will be provided with a 8 question patient survey to complete and return, as well as a food diary that they will complete over a 3 day period to assess their average caloric intake.

SUMMARY:
The goal of this study is to observe the impact of caloric intake on ovarian reserve as measured by anti-müllerian hormone (AMH) levels and antral follicles (AFC) visualized on ultrasound. It has been shown that obesity negatively impacts these markers, but research is lacking regarding the influence of nutrition and caloric intake on fertility. This would give the investigators information on how diet may impact ovarian reserve in patients seeking fertility treatment.

DETAILED DESCRIPTION:
Obesity has been linked to poorer quality oocytes, fewer embryos, and poorer outcomes with pregnancy rates and live birth rates when compared to normal BMI patients. Animal and human studies have shown that short term caloric restriction has lead to improved oocyte quality. Clearly obesity has a negative effect on egg quality. Is this related to the caloric quantity that these patients are consuming when compared with normal BMI patients? If caloric quantity has an impact on egg quality and quantity, then more accurate nutritional guidance could be provided to obese patients who desire to undergo fertility treatments to achieve pregnancy. This could ultimately lead to an improvement in pregnancy rates and live birth rates for these patients.

The goal is to create a survey that would ask patients questions about their caloric intake and activity level. They would also be provided with a food diary to track their caloric intake over a three-day period. They will be instructed to complete the diary during a three day period that would represent their typical diet without any modifications or deviations. The investigators would take the information from this survey to look at average daily caloric intake for a single patient. This data would then be compared with AMH (anti-müllerian hormone) levels and antral follicle counts (AFC) seen on US that would be accessible through the patient's chart. This data would be readily accessible as it is part of all patients' initial workup for infertility assessment and treatment. The investigators would allow for up to a 12 month time period between when these lab and ultrasound findings were performed and when the patient is enrolled in the research study in order to accurately reflect patients' average caloric intake.

Antral follicles are visualized and measured by transvaginal ultrasound and defined as measuring 2-10mm in diameter. This study would define a low AFC ranging from 0-10 antral follicles seen between days two and four of a regular menstrual cycle and would be consistent with poor ovarian reserve. AMH is a hormone level that is expressed by early follicles and reflects the size of the follicle pool. This level represents ovarian function and provides additional information on ovarian reserve. This level can be measured anytime during the menstrual cycle. Normal and abnormal values for the AMH lab value will be determined in this study by the specific laboratory assay that is used by Trihealth, and what that laboratory's reference ranges are since there is not an accepted standardized range.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 who are seeking fertility treatment at Bethesda Fertility Center will be included.

Exclusion Criteria:

* Women who have a diagnosis of PCOS will be excluded from the study due to their abnormal AMH and follicle numbers.
* Women will be excluded if more than 12 months has passed since AMH and AFC levels have been measured.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women aged 18-45 who are seeking fertility treatment at the Bethesda Fertility Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Average Daily Caloric Intake | 3 days
  Patients will complete a food diary that they will complete over a 3 day period to assess their average caloric intake.

CONTACTS AND LOCATIONS:
Overall Officials: Kasey Reynolds, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- Bethesda Fertility Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No